CLINICAL TRIAL: NCT02256124
Title: The Effect of Lamotrigine on Cognitive Deficits Associated With Neurofibromatosis Type 1: a Phase II Randomized Controlled Multi-centre Trial (NF1-EXCEL)
Brief Title: Effect of Lamotrigine on Cognition in NF1
Acronym: NF1-EXCEL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to our experience, the small number of new inclusions, and the uncertainty regarding the COVID-19 outbreak, we have decided to discontinue the study.
Sponsor: Erasmus Medical Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, M.J. Ottenhoff, MD, MD, MSc, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC-2013-460; 2013-003405-26 (EudraCT Number); NL 44912.078.13 (Other: The Central Committee on Research Involving Human Subjects (CCMO)); 113303003 (Other Grant/Funding Number: ZonMw, Netherlands Organisation for Health Research and Development)
Record Dates: First submitted 2014-09-17; First posted 2014-10-03 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis type 1; NF1; Cognition; Learning problems; Lamotrigine; Transcranial magnetic stimulation; TMS
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine (Experimental): Lamotrigine during 28 consecutive weeks:
  * 8 weeks dose-increase phase: from 25mg once daily to 100mg twice daily
  * 18 weeks target-dose phase: 100mg twice daily
  * 2 weeks decline-phase: 100mg once daily.
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Placebo tablets during 28 consecutive weeks, with identical appearance to lamotrigine tablets, mimicking the lamotrigine dosing schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine
  Other Names: Lamictal
  Arms: Lamotrigine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether lamotrigine can improve cognitive and neurophysiological deficits in adolescents with Neurofibromatosis type 1.

DETAILED DESCRIPTION:
Cognitive deficits in the autosomal dominant disorder Neurofibromatosis type 1 (NF1) typically consist of a lower than average IQ, impaired visual-spatial learning, attention problems and impaired executive functioning. These deficits have a substantial influence on the daily life of pediatric and adolescent individuals with NF1. One of the key underlying mechanisms of these deficits is an increased gamma-aminobutyric acid (GABA)-ergic inhibition and a subsequent decrease in synaptic plasticity. The ENCORE laboratory has recently shown that loss of the NF1-gene is associated with attenuated function of the hyperpolarization-activated cyclic nucleotide-gated channel 1 (HCN1). These channels, enriched in membranes of inhibitory interneurons, play an important role in the pathophysiology underlying the cognitive deficits in NF1. Lamotrigine, an HCN-agonist, restored function of HCN1, together with the electrophysiological and visual-spatial learning deficits in Nf1-mice. Thus, lamotrigine is a novel candidate drug for treating cognitive deficits associated with NF1.

ELIGIBILITY:
Inclusion Criteria:

* NF1 patients with a genetically confirmed diagnosis
* Age 12-17.5 years at inclusion
* Oral and written informed consent by parents and assent from participants

Exclusion Criteria:

* Segmental NF1
* Severe hearing problems or deafness
* Severe visual problems or blindness
* Use of the following medication, as of interaction with lamotrigine: phenytoin, carbamazepine, phenobarbital, primidon, rifampicin, atazanavir/ritonavir, lopinavir/ritonavir, oxcarbazepine, topiramate, oral contraceptive pill including stop-week (estrogen and progesterone) and valproic acid during 3 months before inclusion.
* Use of psycho-active medication other than methylphenidate
* Previous allergic reactions to anti-epileptic drugs
* Epilepsy or epilepsy in the past
* Suicidal thoughts or behaviour
* Renal insufficiency
* Liver insufficiency
* Pregnancy
* Brain tumour or other brain pathology potentially influencing the outcome measures

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Performance intelligence quotient (change from baseline) | Baseline and 26 weeks
  Assessed by the Wechsler Intelligence Scales for Children - third edition (WISC-III).

SECONDARY OUTCOMES:
Visual-spatial working memory (change from baseline) | Baseline and 26 weeks
  Assessed by the Paired Associative Learning (PAL) task of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
Visual perception (change from baseline) | Baseline and 26 weeks
  Assessed by the Motor Free Visual Perception Test - third edition (MVPT-3).
Sustained attention (change from baseline) | Baseline and 26 weeks
  Assessed by the Sustained Attention DOTS (SA-DOTS) of the Amsterdam Neuropsychological Tasks (ANT).
Visual-motor integration (change from baseline) | Baseline and 26 weeks
  Assessed by the Beery-Buktenica Developmental Task of Visual Motor Integration - sixth edition (Beery-VMI-6).
Fine motor coordination (change from baseline) | Baseline and 26 weeks
  Assessed by the Grooved Pegboard Test.
Attention problems (change from baseline) | Baseline, 10 weeks, 26 weeks and 52 weeks
  Assessed by a parent rated ADHD-questionnaire, the ADHD-vragenlijst (AVL).
Executive functioning (change from baseline) | Baseline, 26 weeks and 52 weeks
  Assessed by the Behavior Rating Inventory for Executive Function parent questionnaire (BRIEF).
Short intracortical inhibition (SICI) (change from baseline) | Baseline and 10 weeks
  Assessed by paired pulse transcranial magnetic stimulation (ppTMS).
Long-term potentiation-like plasticity (change from baseline) | Baseline and 10 weeks
  Assessed by paired associative stimulation (PAS) using transcranial magnetic stimulation (TMS).

OTHER OUTCOMES:
Full IQ (Intelligence Quotient) | Baseline
  Assessed by the Wechsler Intelligence Scales for children - third edition (WISC-III).
Adverse event registration | Baseline, 4 weeks, 8 weeks, 10 weeks, 14 weeks, 18 weeks, 26 weeks, 28 weeks and additionally on indication
NF1 disease severity | Baseline
  Assessed by the Riccardi scale.
Physical examination | Baseline, 10 weeks and 26 weeks
Pharmacokinetics: Area under the curve (AUC) and average steady state concentration. | 10 weeks, 18 weeks and 26 weeks
  Pharmacokinetic model build with NONMEM analysis of trough level, Tmax level and a level 6 hours post-dose.
Kidney function | Baseline and 10 weeks
  Urea, creatinine
Hepatic enzymes | Baseline and 10 weeks
  ALAT, ASAT, GGT
Full blood count | Baseline and 10 weeks
Parental education | Baseline
  Determined by highest educational grade as measured with the "Standaard Onderwijsindeling (SOI)" classification by Statistics Netherlands (Centraal Bureau voor Statistiek; CBS)
Parental occupation | Baseline
  Determined by the most appropriate level of education for the particular occupation
Educational level | Baseline and 26 weeks
  Determined using the ISCED (International Standard Classification of Education) 2011 levels

CONTACTS AND LOCATIONS:
Overall Officials: Ype Elgersma, PhD, Principal Investigator — Erasmus Medical Center; Henriette A Moll, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- University Hospital Leuven, Leuven, Belgium
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Hospital Sant Joan de Deu, Barcelona, Spain

REFERENCES:
- [Derived] Ottenhoff MJ, Heuvelmans A, Castricum J, Tulen JH, Rens G, Fujiyama H, Levin O, Swinnen SP, Moll HA, Wit MY, Elgersma Y. The effect of lamotrigine on cortical inhibition and plasticity in Neurofibromatosis type 1: Exploratory analysis of a randomized controlled trial (NF1-EXCEL). Clin Neurophysiol. 2025 May;173:150-162. doi: 10.1016/j.clinph.2025.02.270. Epub 2025 Mar 10. PMID 40121838
- [Derived] Ottenhoff MJ, Mous SE, Castricum J, Rietman AB, Oostenbrink R, van der Vaart T, Tulen JHM, Parra A, Ramos FJ, Legius E, Moll HA, Elgersma Y, de Wit MY; ENCORE Expertise Center for NF1. Lamotrigine for cognitive deficits associated with neurofibromatosis type 1: A phase II randomized placebo-controlled trial. Dev Med Child Neurol. 2025 Apr;67(4):537-549. doi: 10.1111/dmcn.16094. Epub 2024 Sep 28. PMID 39340758
- See also: ENCORE expertise center — https://www.erasmusmc.nl/nl-nl/sophia/patientenzorg/centra/encore